CLINICAL TRIAL: NCT06243042
Title: A Comparative Study of Vitamin D Serum Levels in Monosymptomatic Enuretic Children and Non-enuretic Children
Brief Title: Vitamin D Serum Levels in Monosymptomatic Enuretic and Non Enuretic Children
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaa Mostafa, Associate Professor, Ain Shams University
Other Study IDs: ASU-7122021
Record Dates: First submitted 2024-01-04; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Nocturnal Enuresis
Keywords: Nocturnal enuresis; Vitamin D
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enuretic: Children complaining of monosymptomatic enuresis
  Interventions: Diagnostic Test: serum vitamin D; Diagnostic Test: urine osmolality; Other: Frequency volume chart
- Non-enuretic: Healthy non enuretic children
  Interventions: Diagnostic Test: serum vitamin D; Diagnostic Test: urine osmolality; Other: Frequency volume chart

INTERVENTIONS:
Diagnostic Test: serum vitamin D — blood sample for serum vitamin D level Vitamin D serum level was measures using the ELISA technique. The Cal Biotech Vitamin D Kit (Mannheim, Germany) was used, which is a solid phase enzyme linked immunoassay (ELISA), based on the principal of competitive binding. Vitamin D deficiency was defined as serum Vit. D below 20 ng/ml.
Diagnostic Test: urine osmolality — nocturnal urine osmolality: Clear instructions for mothers were to let the child void before sleep and every two hours till 8 am. Short intervals were meant to avoid enuretic episodes during calculation of nocturnal urine volume, and if occurred it mandates the repeat of chart on another day.
  Nocturnal urine collected over the night was tested for osmolality, it was measured in mOsm/kg.
Other: Frequency volume chart — volume and frequency from time of sleep till 8 am

SUMMARY:
We are group of researchers interested in causes and management of nocturnal enuresis, we embarked on this research on 2020 and we reached promising results regarding the role of vitamin D serum level in etiology and management of monosymptomatic enuresis.

DETAILED DESCRIPTION:
this research was conducted as a comparative study regarding serum vitamin D levels in monosymptomatic enuretic and non enuretic children, also we compared urine osmolality and nocturnal polyuria in both groups and we found that low vitamin D levels are correlated with low nocturnal urine osmolality and increased incidence of nocturnal polyuria

ELIGIBILITY:
Inclusion Criteria:

* Patients with PMNE.
* which was defined as bedwetting frequency of 3 or more nights per week for at least 2 weeks of observation.
* Didn't receive any previous treatment for enuresis.

Exclusion Criteria:

* Patients with non-monosymptomatic enuresis (associated with storage and/or voiding symptoms). -Patients with anatomical abnormalities (Meatal stenosis, Hypospadias, Epispadias, etc.).
* Patients with neurological diseases.
* Patients with Renal impairment.
* Patient with previous pelvic, urological or brain and spinal cord surgery.
* Patients with chronic constipation and irritable bowel habits.
* Patients with active urinary tract infection.
* Patients who are on vitamin D supplements.

Ages: 5 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: male and female children from 5-15 years wer selcted in two groups 60 enuretic children 60 non enuretic children as a control group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Vitamin D level | through study completion, average 1 year.
  low vitamin d levels in enuretic group

SECONDARY OUTCOMES:
nocturnal polyuria | through study completion, average 1 year.
  frequency volume chart idobtained
low nocturnal urine osmolality | through study completion, average 1 year.
  nocturnal urine osmolality

CONTACTS AND LOCATIONS:
Overall Officials: diaa mostafa, MD, Principal Investigator — Ain Shams University
Locations (1):
- Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mostafa D, Shaker H, Badr A, Abuelnaga M. A Comparative Study of Vitamin D Serum Levels in Monosymptomatic Enuretic Children and Non-Enuretic Children. Neurourol Urodyn. 2025 Jan;44(1):212-219. doi: 10.1002/nau.25618. Epub 2024 Oct 30. PMID 39473396

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT06243042/Prot_SAP_000.pdf